CLINICAL TRIAL: NCT06697093
Title: Polish Nationwide Registry of Diagnostics, Treatment and Outcome in Patients With Cardiogenic Shock CaS-POL
Brief Title: Polish Nationwide Registry of Diagnostics, Treatment and Outcome in Patients With Cardiogenic Shock
Acronym: CaS-POL
Status: Recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Collaborators: Polish Cardiac Society (Other); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Wiktor Kuliczkowski, MD, PhD, Associate Professor, Head of the Catheterization Laboratory at Wroclaw University Hospital, Wroclaw Medical University
Other Study IDs: KB/16/2023/N
Record Dates: First submitted 2024-11-06; First posted 2024-11-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock
Keywords: mechanical circulatory support; myocardial infarction; Cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- cardiogenic shock patients: The registry will include all patients presenting with primary cardiogenic shock. All medical interventions will be conducted based on established clinical indications.

SUMMARY:
The registry objective is to get information on current epidemiology, diagnostics, treatment and outcome in patients with cardiogenic shock in Poland. Obtained information will help to plan the nationwide initiative for modern cardiogenic shock treatment with established place for mechanical circulatory support.

It is hypothesized that the treatment and outcome of cardiogenic shock, including mechanical circulatory support, are currently poor in Poland and should be improved. Unfortunately, without status quo data, efficient planning for its improvement cannot be conducted, hence the CaS-POL registry initiative.

DETAILED DESCRIPTION:
The prospective registry will be open in nature; any cardiology department in Poland with access to a 24-hour hemodynamic laboratory will be eligible to participate in the study. All participants will use an electronic CRF (Case Report Form) to anonymously collect data on the incidence, etiology, diagnosis, treatment approaches, and prognosis of patients with cardiogenic shock. Data will be collected by researchers from the medical documentation of participating centers. The data collection period will span six months, followed by a six-month prospective observation through visit in person, per telephone contact to the patient or his/her relatives or by retracting National Health Fund data in case the contact to the patient or his/her relatives is impossible.

To enable comparison with global data, collected information will include, among other aspects, the latest Society for Cardiovascular Angiography and Interventions (SCAI) classification for cardiogenic shock, the availability and application of modern short- and long-term mechanical circulatory support techniques, and the frequency of heart transplants.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock patients of all etiologies in SCAI stage B, C, D, E.
* age > 18 years old
* persistent hemodynamic failure defined as systolic blood pressure of <90 mmHg for ≥ 30 minutes or the requirement for inotropic or vasopressor agents with evidence of hypoperfusion of the peripheral organs

Exclusion Criteria:

* patients without return of spontaneous circulation who were considered to extracorporeal cardiopulmonary resuscitation (ECPR)
* primary septic, anaphylactic, hypovolemic shock
* post-operative cardiogenic shock
* end-stage of heart failure disqualified from mechanical circulatory support and heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Unit (ICU) in the Cardiology, Cardiac Surgery, or to the Anesthesiology departments with a clinically evident cardiac etiology of shock.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | From the date of cardiogenic shock diagnosis recognition until the date of death from any cause assessed up to 6 months
  all-cause mortality

SECONDARY OUTCOMES:
myocardial infarction | From the date of cardiogenic shock diagnosis recognition until the date of first documented myocardial infarction assessed up to 6 months
  Recurrent myocardial infarction following an initial event
stroke | From the date of cardiogenic shock diagnosis recognition until the date of first documented stroke assessed up to 6 months
  stroke following an initial event
heart transplantation | From the date of cardiogenic shock diagnosis recognition until the date of heart transplantation assessed up to 6 months
  Heart transplantation in patients without myocardial recovery following cardiogenic shock.
long-term LVAD implantation | From the date of cardiogenic shock diagnosis recognition until the date of long-term LVAD assessed up to 6 months
  Long-term LVAD implantation in patients without myocardial recovery following cardiogenic shock

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Institute of Heart Diseases, Wroclaw Medical University, Wroclaw, Poland, Wroclaw, Lower Silesian Voivodeship
  - Wroclaw Medical University, Wroclaw

IPD SHARING:
Plan to Share IPD: No